CLINICAL TRIAL: NCT06411886
Title: Optimizing the Measurement of Therapeutic Targets for Treatment of Asthma Induced by Allergen Inhalation Challenge in Mild Allergic Asthma
Brief Title: Measurements of Inflammation Induced by Allergen Inhalation Challenge in Mild Allergic Asthma
Acronym: MATT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Principal Investigator, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MATT-17085
Record Dates: First submitted 2024-03-11; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Mild Asthma
MeSH Terms: interventions — Bronchial Provocation Tests

STUDY DESIGN:
Intervention Model Description: Randomized placebo control two way crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergen Challenge (Experimental): Inhaled allergen
  Interventions: Diagnostic Test: Allergen challenge
- Diluent Challenge (Placebo Comparator): Inhaled saline
  Interventions: Diagnostic Test: Saline challenge

INTERVENTIONS:
Diagnostic Test: Allergen challenge — Inhaled allergen
  Arms: Allergen Challenge
Diagnostic Test: Saline challenge — Inhaled saline
  Arms: Diluent Challenge

SUMMARY:
This study will measure lung function tests and examine biological samples collected before and after inhaled allergen challenges and diluent (control) challenges in participants with mild allergic asthma.

DETAILED DESCRIPTION:
This study will measure lung function tests examine biological samples collected before and after inhaled allergen challenges and diluent (control) challenges in participants with mild allergic asthma. Each inhaled challenge will consist of 3 consecutive days (triads) where participants will inhale either allergen extract or saline diluent (control) and airway function will be measured, and biological samples will be obtained. Inhaled allergen challenges will be controlled, with diluent inhalation challenge in a randomized crossover design. Each participant will be required to attend the research lab on at least three consecutive days for an inhaled challenge triad. On triad Day 1, study staff will provide an overview of the study purpose and procedure and answer any questions the participant may have. The individual will then provide informed consent if they wish to participate (i.e. sign the consent form), and safety labs will be collected for blood chemistry and hematology, urinalysis. Skin prick testing will be conducted to determine relevant allergen sensitivities and to determine which allergen extract will be used for the skin test titration and inhalation. A pre-allergen challenge methacholine test is conducted, followed by sputum induction, blood draw and nasal brushing. On Day 2 of the triad, the participant will inhale a dose of allergen that is 3 doubling doses lower than that estimated (using methacholine test and skin titration) to give a 20% fall in forced expiratory volume in 1 second. The participant will continue inhaling doubling doses of allergen extract until a 20% fall in forced expiratory volume in 1 second has been reached. Spirometry will be performed for 7 hours. At 7h post-inhalation a bronchodilator will be administered, and a sputum sample will be collected. Participants will be sent home with bronchodilator to use if needed. On Day 3 of the triad, participants will return at approximately 24h post-allergen challenge for a methacholine test, sputum induction, blood draw and nasal brushing.

Participants will also undergo a Triad 2 (Days 1-3) for an inhaled challenge with 0.9% saline. The intervention (allergen or diluent) will be randomized to Triad 1 or Triad 2. A four-week washout is required between allergen inhalation and a subsequent diluent inhalation. A one-week washout is required between diluent inhalation and a subsequent allergen inhalation.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged 18 to 75 years inclusive at the first screening visit with mild atopic asthma.

General good health with no other medical condition, medication use or lifestyle activities that would influence the outcome of the allergen challenge (case by case, investigator discretion)

A forced expiratory volume after 1 second greater than 70% predicted at the first screening visit.

A methacholine provocative concentration causing a 20% fall in forced expiratory volume in 1 second of ≤ 16 mg/ml during the first methacholine inhalation challenge.

Positive skin test to at least one common aeroallergen.

A demonstrated (or historic documentation of) early asthmatic response following the allergen inhalation challenge.

Agree to withhold use of inhaled short-acting β2-agonist for 8 hours before all study visits where spirometry is performed.

Agree to refrain from rigorous exercise 4 hours before all study visits.

Nonsmoker or former smoker (former smokers are permitted if nonsmoker for 2 years and <10 pack-year smoking history).

Capable of performing the maneuvers and procedures required by the protocol and have a high probability for compliance with and completion of the study.

Exclusion Criteria:

Upper or lower respiratory infection or asthma exacerbation within 4 weeks of first study visit. The occurrence of allergic rhinitis, as determined by investigator, will not exclude the subject from the study.

Use of any medications for treatment of asthma other than prophylactic short-acting β2-agonists, or intermittent (not more than once weekly) use of short-acting β2-agonists for relief of symptoms.

Current or history of lung disease other than mild stable allergic asthma. Smoking within past 12 months, or former smoker with >10-pack-year history.

Known to have tested positive for human immunodeficiency virus or hepatitis. For women only - self-reported pregnancy, breast-feeding, or plans to become pregnant during the study.

Reported use of illegal drugs or history of abuse of prescription drugs or alcohol within 1 year before the first screening visit.

Any clinically important deviation from normal limits in vital signs.

Participation in a research study with an investigational product during the last 30 days or 5 half-lives of the drug (whichever is longer) Inability to produce a sputum sample at the first study visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 | 7 hours post-allergen challenge
  FEV1 after allergen challenge expressed as a percentage of the pre-allergen baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario